CLINICAL TRIAL: NCT04041687
Title: Outpatient Cervical Ripening with Misoprostol in Low-Risk Inductions After 39 Weeks Gestation: a Cost, Safety, and Satisfaction Analysis
Brief Title: Outpatient Cervical Ripening
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: pro00084666
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy
Keywords: induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The process of labor induction can mean several hours or even days spent as an inpatient prior to delivery. These prolonged hospital admissions contribute to increased financial burden on both patients and hospital systems, dissatisfaction with induction length, and staffing concerns. Several obstetric practices in the U.S. have already incorporated outpatient cervical ripening (the beginning of the induction process) into their regular practices. The investigators aim to determine if outpatient cervical ripening is a safe, non-inferior, and preferred option to the traditional inpatient induction process.

DETAILED DESCRIPTION:
This study will attempt to assess whether outpatient cervical ripening with misoprostol, a synthetic PGE1 analog (Cytotec(R), Pfizer), is an effective and safe option for low-risk pregnant women at or after 39 weeks gestation with an unfavorable cervix. This study comes in the wake of the ARRIVE trial, which may reasonably increase the number of low-risk term inductions.

The process of labor induction, including cervical ripening, can take several hours or even days. This prolonged course contributes not only to long hospital stays and subsequently increased financial burden to both patients and healthcare systems, but also to patient and provider dissatisfaction with length of induction. Additionally, with the expected increase in elective inductions of primigravid women with unfavorable cervices as a result of the ARRIVE study, hospitals face the possibility of being at capacity on labor and delivery with inadequate staffing to ensure patient safety.

Traditionally, the process of cervical ripening begins after inpatient hospital admission. Several small studies have evaluated outpatient ripening with various agents including foley balloon catheters, PGE1 analogs such as misoprostol, and other prostaglandins. The American College of Obstetricians and Gynecologists has commented on the limited data available on outpatient cervical ripening safety and efficacy, noting that outpatient cervical ripening is "appropriate for carefully selected patients" in Practice Bulletin 107. Data have been reassuring as far as safety and efficacy based on several studies, but are limited due to small sample size, For example, a randomized, double-blind placebo-controlled study in 2009 found that outpatient oral misoprostol for late term pregnancies had a significantly shorter time from study entry to spontaneous labor and delivery. This study showed no difference in fetal or maternal morbidity, but was not powered to safety as there were only 44 subjects per group (10). Some institutions including OB/GYN groups at Beth Israel Deaconess Hospital, South Shore Hospital in MA, and Alaska Native medical center have incorporated outpatient ripening into their everyday practices, but little data on outcomes have been published from these sites.

The investigators aim to determine if outpatient cervical ripening is a safe, non-inferior option to the traditional inpatient cervical ripening. The investigators will evaluate whether outpatient ripening impacts patient satisfaction, patient/hospital costs, and adverse outcomes in our health system setting. Cervical ripening is standard care at other OB/GYN practices across the county and the investigators intend to apply this care pathway for patients. The investigator's goal is to ensure the safety of participants by carefully selecting low risk patients and providing necessary fetal monitoring before and after administration. The results of this study can be used to determine if outpatient cervical ripening can be incorporated in daily practices of OB/GYN providers at GHS.

ELIGIBILITY:
Inclusion Criteria:

* Low risk, pregnant women seeking elective induction of labor after 39 weeks gestation
* Women without a medical indication for induction of labor.
* Multigravida or primigravida women who are scheduled for late term (postdates) induction will be included.

Exclusion Criteria:

* Previous cesarean section,
* Any contraindication to labor or vaginal delivery,
* A ny patients where misoprostol should be used with caution (IUGR, oligohydramnios)
* Bishop score > 6
* ruptured amnioticmembranes

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnancy is condition of gender
Study Population: Low risk pregnant womenn
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Assess outpatient cervical ripening protocol feasibility | one year
  length of induction misoprostol, a synthetic PGE1 analog (Cytotec®, Pfizer, New York), is an effective and safe option for low-risk pregnant women with an unfavorable cervix at or after 39 weeks gestation.
Assess outpatient cervical ripening protocol feasibility | one year
  unplanned/unanticipated admissions
Assess outpatient cervical ripening protocol feasibility | one year
  Rate of change in Bishop score
Assess outpatient cervical ripening protocol feasibility | one year
  number of misoprostol doses required
Assess outpatient cervical ripening protocol feasibility | one year
  number of cervical checks performed
Assess outpatient cervical ripening protocol feasibility | one year
  rates of chorioamnionitis or endometritis
Assess outpatient cervical ripening protocol feasibility | one year
  fetal or neonatal complications
Assess outpatient cervical ripening protocol feasibility | one year
  other maternal complications of induction or delivery
Assess outpatient cervical ripening protocol feasibility | one year
  apgar scores
Assess outpatient cervical ripening protocol feasibility | one year
  route of delivery - vaginal delivery with or without assistance, cesarean section and indication
Assess outpatient cervical ripening protocol feasibility | one year
  satisfaction - patient and provider, via survey (labor agentry questionnaire) for outpatient group

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Demosthenes, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No